CLINICAL TRIAL: NCT00004796
Title: Phase II Study of Lactulose and Circadian Rhythms in Patients With Cirrhosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Northwestern University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/11934; NU-523
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-02

CONDITIONS: Portal Hypertension; Hepatic Encephalopathy; Cirrhosis
Keywords: cardiovascular and respiratory diseases; cirrhosis; gastrointestinal disorders; hypertensive disorder; portal hypertension; rare disease
MeSH Terms: conditions — Hypertension, Portal; Hepatic Encephalopathy; Fibrosis; Respiratory Tract Diseases; Gastrointestinal Diseases; Hypertension; Rare Diseases | interventions — Lactulose

INTERVENTIONS:
Drug: lactulose

SUMMARY:
OBJECTIVES: I. Assess the effect of lactulose on the circadian rhythm of plasma melatonin in patients with subclinical hepatic encephalopathy.

II. Assess the intrasubject variability of circadian melatonin levels and neuropsychological tests.

III. Assess which elements of the neuropsychological test battery show the response to lactulose.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients are alternately assigned to 1 of 2 treatment groups: no therapy for 3 weeks followed by lactulose for 3 weeks versus lactulose for 3 weeks followed by no therapy for 3 weeks.

A dietician advises patients on a 1 g/kg per day protein diet. The lactulose dose is adjusted to result in 2 or 3 loose bowel movements per day.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Clinical diagnosis of cirrhosis with portal hypertension or portal-systemic shunting

--Prior/Concurrent Therapy--

* No concurrent therapy for hepatic encephalopathy

--Patient Characteristics--

* Age: Under 65
* Performance status: Not specified
* Hematopoietic: Not specified
* Hepatic: See Disease Characteristics
* Renal: Not specified
* Other: No alcohol intake within 1 month prior to entry No requirement for beta blockers No requirement for corticosteroids Not in intercontinental travel

Ages: 0 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16
Dates: Start 1994-11; Study Completion 1997-02

CONTACTS AND LOCATIONS:
Overall Officials: Andres Blei, Study Chair — Northwestern University